CLINICAL TRIAL: NCT00753207
Title: An Open-Label Phase I Study of Fixed Dose Lapatinib in Combination With an Escalating Dose of Epirubicin in Metastatic Breast Cancer
Brief Title: Lapatinib and Epirubicin in Treating Patients With Metastatic Breast Cancer. ICORG 06-30
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-30 ICORG; ICORG-06-30; ICORG-109403; EUDRACT-2007-002327-33; EU-20875; NCT00566748 (obsolete NCT alias)
Record Dates: First submitted 2008-09-13; First posted 2008-09-16 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2014-01

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Lapatinib; Immunohistochemistry; Chromatography, Liquid; Mass Spectrometry

ARMS (1):
- Lapatinib and Epirubicin (Experimental): Fixed dose of lapatinib in combination with escalating dose of epirubicin.
  Interventions: Drug: epirubicin hydrochloride; Drug: lapatinib ditosylate; Other: biomarker analysis; Other: immunohistochemistry staining method; Other: liquid chromatography; Other: mass spectrometry

INTERVENTIONS:
Drug: epirubicin hydrochloride
Drug: lapatinib ditosylate
Other: biomarker analysis
Other: immunohistochemistry staining method
Other: liquid chromatography
Other: mass spectrometry

SUMMARY:
RATIONALE: Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as epirubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving lapatinib together with epirubicin may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of epirubicin when given together with lapatinib in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the safety and tolerability of fixed-dose lapatinib ditosylate in combination with epirubicin hydrochloride in patients with metastatic breast cancer.
* To determine the optimally-tolerated regimen in these patients.

Secondary

* To determine the clinical efficacy of this regimen in these patients.
* To analyze pharmacokinetic data of this regimen.
* To determine biomarkers that correlate with clinical benefit or response to lapatinib ditosylate in these patients.

Tertiary

* To identify tumor-derived or blood-derived biomarkers that correlate with or are predictive of clinical response or benefit to lapatinib ditosylate in these patients.
* To determine the levels of IGF-IR and phosphorylated IGF-IR in tumor tissue.
* To determine the expression pattern of the proteins associated with drug resistance that may be clinically active in these patients.

OUTLINE: This is a multicenter, dose-escalation study of epirubicin hydrochloride.

Patients receive oral lapatinib ditosylate followed by epirubicin hydrochloride IV over 15-30 minutes on day 1. Treatment repeats every 3 weeks for up to 7 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for pharmacokinetic analysis via liquid chromatography-mass spectometry (LC-MS).

After completion of study therapy, patients are followed at 28 days and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of breast cancer

  * Metastatic disease
* No de novo metastasis
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy > 3 months
* Menopausal status not specified
* ANC ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 9 g/dL
* Creatinine clearance ≥ 50 mL/min
* AST/ALT < 3 times upper limit of the normal (ULN)
* Total bilirubin normal (unless documented history of congenital hypobilirubinemia)
* LVEF normal by ECHO or MUGA scan
* Not pregnant or breastfeeding
* Negative pregnancy test
* Fertile patients must use effective contraception from the time of their negative pregnancy test before treatment, during treatment, and 28 days following treatment
* Able to swallow and retain oral medication
* History of other malignancies (e.g., cervical carcinoma in situ, melanoma in situ, or basal cell or squamous cell carcinoma of the skin) allowed provided patient has been treated and disease free ≥ 5 years and deemed by the investigator to be at low risk for recurrence
* No known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to lapatinib ditosylate or excipients
* No malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach or small bowel, or ulcerative colitis
* No active or uncontrolled infection
* No known history of uncontrolled or symptomatic angina, arrhythmias, congestive heart failure, or other cardiac disorders
* No history of prolonged QT interval
* No active hepatic or biliary disease (except for Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* No concurrent disease or condition that would render the patient inappropriate for study participation, or serious medical disorder that would interfere with the patient's safety
* No dementia, altered mental status, or psychiatric condition that would prohibit the understanding or rendering of informed consent

PRIOR CONCURRENT THERAPY:

* Prior radiotherapy for treatment of primary tumor allowed
* Prior non-anthracycline based regimens in neoadjuvant, adjuvant, or metastatic setting allowed
* Prior adjuvant Herceptin® or ErbB inhibitors allowed provided disease progression was > 6 months after completion of treatment
* More than 3 months since prior Herceptin®, ErbB1, or ErbB2
* No prior chemotherapy in the adjuvant or neoadjuvant setting with anthracycline or anthracenedione-containing regimens
* More than 3 weeks since prior and no concurrent medications that would prolong QT interval
* More than 1 month or 5 half-lives (whichever is longer) since prior, no concurrent investigational drugs
* No unresolved or unstable, serious toxicity from prior investigational drug and/or cancer treatment
* At least 3 weeks since prior and no concurrent prohibited medications (i.e., CYP3A4 inducers or inhibitors)
* No concurrent non-study anticancer therapy (i.e., chemotherapy, immunotherapy, or biologic therapy)
* No concurrent participation in another clinical trial
* No concurrent grapefruit or grapefruit juice
* Concurrent bisphosphonates allowed

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-10; Primary Completion 2008-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Optimally-tolerated regimen of lapatinib ditosylate in combination with epirubicin hydrochloride | 2012

SECONDARY OUTCOMES:
Efficacy of this regimen in terms of objective tumor response rate and disease progression as assessed by standard RECIST criteria | 2012
Pharmacokinetics | 2012
Correlation between baseline expression of intra-tumoral biomarkers (e.g., ErbB1, ErbB2, insulin-like growth factor-1 receptor, p-AKT, and ERK) and clinical response or benefit to lapatinib ditosylate by IHC | 2012
Correlation between expression pattern of drug resistance proteins (e.g., p-glycoprotein, MRP1, BCRP, and MDR-3) and clinical response or benefit to lapatinib ditosylate by IHC | 2012

CONTACTS AND LOCATIONS:
Overall Officials: John Crown, MD, Principal Investigator — St Vincent's University Hospital, Ireland
Locations (3):
- Ireland (3):
  - The Adelaide and Meath Hospital, Dublin Incorporating the National Childresn's Hospital, Dublin
  - St Vincent's University Hospital, Dublin
  - St James's Hospital, Dublin